CLINICAL TRIAL: NCT01080937
Title: French Observatory of Acute Heart Failure
Acronym: OFICA
Status: Completed | Type: Observational
Sponsor: French Cardiology Society (Other)
Responsible Party: Sponsor
Other Study IDs: SFC-OFICA
Record Dates: First submitted 2010-03-01; First posted 2010-03-05 (Estimated); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Acute Heart Failure
Keywords: acute heart failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patient with acute heart failure: Hospitalized patient, whatever the mode of initial admission with acute heart failure

SUMMARY:
During the last decade, progress has been made in the management of heart failure. However, the changing characteristics of patients and practices in the "real world" and their impact on the prognosis of patients admitted for acute heart failure remain poorly studied.

2000 consecutive patients recruited in a single day in hospitals volunteered to participate in the cohort during a day dedicated.

DETAILED DESCRIPTION:
The total duration of recruitment is one day (date to be set soon by the Executive Committee): all patients hospitalized, and whatever their date of admission with the diagnosis of heart failure will be selected for the study.

Information on each hospital stay will be obtained at baseline and at the end of the hospitalization by the hospital teams.

A telephone follow-up will be conducted at 3 months among survivors and / or their doctor by CRAs dedicated to the French Society of Cardiology.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age (e) over 18 years
2. Inpatient, whatever the mode of initial admission with acute heart failure (de novo heart failure or decompensation of chronic heart failure) regardless of severity, corresponding to one of the following clinical situations (clinical criteria in Appendix 1):

   * Pulmonary edema, hypertensive or not
   * congestive heart failure (pulmonary congestion and peripheral edema)
   * cardiogenic shock
   * Insufficient high output cardiac
3. Patients who agreed to participate in the study
4. Isolated right heart failure

Exclusion Criteria:

1. expressed refusal to participate in the study
2. Hospitalization scheduled for review
3. Background surgery (immediate postoperative period)
4. Diagnosis of acute heart failure reversed in favor of an alternative diagnosis before discharge from hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patient, whatever the mode of initial admission with acute heart failure (de novo heart failure or decompensation of chronic heart failure)
Sampling Method: Non-Probability Sample
Enrollment: 1818 (Actual)
Dates: Start 2009-03; Primary Completion 2010-12 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Survival at 3 months | 3 months
  Analyze survival 3 months after the end of initial hospitalization

SECONDARY OUTCOMES:
Hospital Methods | 3 months
  Compare methods of care based on clinical characteristics and hospital structures.
Patterns of admission | 3 months
  Analyze patterns of admission and discharge of patients, depending on their characteristics
Co-morbidities | 3 months
  Analyze the co-morbidities and their impact on care and survival
Drug treatments | 3 months
  Analyze the evolution of drug treatment between the output and monitoring to 3 months
Resources specific diagnostic | 3 months
  Analyze the use of resources specific diagnostic: measurement of BNP or NTproBNP, conducting echocardiogram, coronary angiography, Holter-ECG, Cardiac MRI, Cardiac CT
Therapeutic resources | 3 months
  Analyze the use of therapeutic resources based on specific clinical features: intensive care, ventilation, inotropes, ultrafiltration, introduction of beta-blockers, stimulation, implantable cardioverter defibrillator, circulatory support, graft
During of stay | 3 months
  Analyze the duration of stay according to clinical characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Damien DL LOGEART, Principal Investigator — French Cardiology Society
Locations (1):
- Lariboisiere Hospital, Paris, France

REFERENCES:
- [Result] Logeart D, Isnard R, Resche-Rigon M, Seronde MF, de Groote P, Jondeau G, Galinier M, Mulak G, Donal E, Delahaye F, Juilliere Y, Damy T, Jourdain P, Bauer F, Eicher JC, Neuder Y, Trochu JN; Heart Failure of the French Society of Cardiology. Current aspects of the spectrum of acute heart failure syndromes in a real-life setting: the OFICA study. Eur J Heart Fail. 2013 Apr;15(4):465-76. doi: 10.1093/eurjhf/hfs189. Epub 2012 Nov 27. PMID 23186936
- [Result] Logeart D. [The OFICA study of acute heart failure]. Soins. 2013 Apr;(774):35. No abstract available. French. PMID 23697057